CLINICAL TRIAL: NCT02382224
Title: Worry Exposure for Generalized Anxiety Disorder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient study staff
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Mark B. Powers, Research Associate Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-02-0025
Record Dates: First submitted 2015-02-07; First posted 2015-03-06 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Generalized Anxiety Disorder
Keywords: generalized anxiety disorder; anxiety; worry exposure; treatment
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders | interventions — glutamate decarboxylase 1; Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Worry Exposure for GAD (Experimental): WE is an optimized protocol that incorporates elements of CBT, without the addition of other miscellaneous methods of treatment. A therapist manual will be used and followed at all times to ensure standardized delivery of the program. Interventions that uniquely focus on addressing GAD symptoms will include confronting physical or imagined stimuli through in vivo exposure and WE respectively. Avoidance behaviors will be monitored and reduced systematically, an outcomes will be assessed at baseline, during the 12-week intervention, and at 6-month follow-up.
  Interventions: Behavioral: Worry Exposure for GAD
- 12-week Waitlist (Placebo Comparator): Those who are randomized to the waitlist condition will wait for 12 weeks before beginning the worry exposure.
  Interventions: Behavioral: 12-week Waitlist

INTERVENTIONS:
Behavioral: Worry Exposure for GAD — WE is an optimized protocol that incorporates elements of CBT, without the addition of other miscellaneous methods of treatment. A therapist manual will be used and followed at all times to ensure standardized delivery of the program. Interventions that uniquely focus on addressing GAD symptoms will include confronting physical or imagined stimuli through in vivo exposure and WE respectively. Avoidance behaviors will be monitored and reduced systematically, an outcomes will be assessed at baseline, during the 12-week intervention, and at 6-month follow-up.
  Arms: Worry Exposure for GAD
Behavioral: 12-week Waitlist — Those who are randomized to the waitlist condition will wait for 12 weeks before beginning the worry exposure.
  Arms: 12-week Waitlist

SUMMARY:
The purpose of this study is to examine the efficacy of a worry exposure intervention, a form of cognitive behavioral therapy (CBT), in comparison to a waitlist condition for the treatment of Generalized Anxiety Disorder. There will be a total of 60 subjects enrolled at the University of Texas at Austin. Patients will be randomized (like a flip of a coin) to either 12-sessions of WE therapy or a 12-week waitlist before being offered entry into therapy.

DETAILED DESCRIPTION:
This application proposes a randomized controlled trial, which aims to examine the efficacy of a worry exposure (WE) intervention for the treatment of generalized anxiety disorder (GAD). This protocol is based on a GAD treatment manual first tested in Germany. It has been translated into English, but this version has not yet been tested.

A growing body of research calls for the development of novel interventions for individuals with GAD. GAD is a chronic and debilitating condition with high rates of recurrence, with a lifetime prevalence of 5.7%. Although efficacious psychological interventions exist, many are either not receiving these interventions or remain highly symptomatic following the termination of these interventions. More specifically, cognitive behavioral therapy (CBT) is the only empirically supported treatment for GAD. However, many patients relapse or continue to experience significant symptoms after treatment. Up to 57% of patients do not meet criteria for high endstate functioning after CBT. Together, these findings call for the development of better interventions that are efficacious and easy to disseminate.

The core symptom of GAD is persistent and uncontrollable worry, which allows the individual a way to cognitively avoid perceived threats and emotionally dangerous situations. One study examined the efficacy of WE alone, applied relaxation (AR) alone, and a WL control group, finding that WE was an effective treatment for GAD, concluding that WE should be developed further. Given other areas of avoidance for patients with GAD, the authors recommended adding in vivo exposure in future trials.

The present application proposes to test WE with the addition of in vivo exposure in the United States as an effective treatment for GAD. The present study involves the randomization of 60 adults with GAD to either (1) 12-sessions of WE therapy or (2) a 12-week waitlist (WL), before entering into therapy. The authors hypothesize that participants in the WE intervention will evidence greater reductions in anxiety symptom severity and measures of quality of life relative to individuals randomized to the WL.

ELIGIBILITY:
Inclusion Criteria:

* be between 18 and 65 years of age
* principal diagnosis of Generalized Anxiety Disorder
* be willing to and capable of providing informed consent, attending all study visits, and complying with the protocol

Exclusion Criteria:

* current diagnosis of a psychotic, developmental, or bipolar disorder
* significant suicide risk as determined by structured interview
* psychoactive substance dependence within the past 3 months
* Inability to communicate in English
* limited mental competency and the inability to give informed, voluntary, written consent to participate
* psychotropic medications are acceptable only if they are stabilized for at least 3 weeks prior to the baseline visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Change in Penn State Worry Questionnaire (PSWQ). | Up to 6 months
  The PSWQ will be administered 6 separate occasions. The investigators will measure the change in PSWQ scores from pre-treatment to weeks 3, 6, 9, 12, and 38. The PSWQ is a 16-item inventory designed to capture the generality, excessiveness, and uncontrollability of pathological worry. It has been shown to have good internal consistency with samples consisting of older adults with GAD, community subjects, and undergraduates. It has also demonstrated good test-retest reliability over 8-10 weeks.

SECONDARY OUTCOMES:
Beck Anxiety Inventory (BAI). | Up to 6 months
  The BAI will be administered 6 separate occasions. The investigators will measure the change in BAI scores from pre-treatment to weeks 3, 6, 9, 12, and 38. The BAI is a commonly used 21-item, self-report inventory designed to measure severity of anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Mark B Powers, Ph.D., Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States